CLINICAL TRIAL: NCT03639363
Title: Study on the Effect of the Universal Decontamination With Daily Bathing With 4% Chlorhexidine Gluconate on the Incidence of Hospital Acquired Infections in Intensive Care Units
Brief Title: 4% Chlorhexidine Gluconate Daily Bathing for Prevention of Hospital-acquired Infections in Intensive Care Settings
Acronym: Duclorexint
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Of Perugia (Other)
Collaborators: Fondazione Toscana Gabriele Monasterio (Other)
Responsible Party: Principal Investigator, Carlo Pallotto, Medical Doctor, Principal investigator, University Of Perugia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Duclorexint
Record Dates: First submitted 2018-08-13; First posted 2018-08-21 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Hospital Infection
Keywords: 4% chlorhexidine gluconate; infection control
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Experimental): daily bathing with 4% chlorhexidine gluconate soap-like solution followed by water rinsing
  Interventions: Drug: 4% chlorhexidine gluconate soap-like solution
- Control Arm (Active Comparator): daily bathing with standard soap
  Interventions: Other: standard soap

INTERVENTIONS:
Drug: 4% chlorhexidine gluconate soap-like solution — 1. humidify the whole body surface with the exception of the face using water-impregnated washcloths
  2. use 4% CHG-impregnated washcloths to bath the whole body surface with the exception of the face; use at least 30 ml of 4% CHG
  3. wait for at least 30 seconds
  4. rinse using water-impregnated washcloths
  Arms: Intervention Arm
Other: standard soap — 1. humidify the whole body surface with the exception of the face using water-impregnated washcloths
  2. use standard soap-impregnated washcloths to bath the whole body surface with the exception of the face
  3. wait for at least 30 seconds
  4. rinse using water-impregnated washcloths
  Arms: Control Arm

SUMMARY:
The study will assess the utility of 4% chlorhexidine gluconate (CHG) daily bathing to reduce hospital acquired infections in patients admitted to intensive care units. One group will be daily bathed with 4% CHG and the other group with standard soap.

ELIGIBILITY:
Inclusion Criteria:

* admission to the intensive care unit (ICU) or to the post-operative cardiosurgical ICU (PC-ICU)
* ICU/PC-ICU stay for at least 1 night

Exclusion Criteria:

* known allergy to chlorhexidine
* burns, toxic epidermal necrolysis or Stevens-Johnson syndrome as admission diagnosis
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 449 (Actual)
Dates: Start 2015-08-10 (Actual); Primary Completion 2016-04-28 (Actual); Study Completion 2016-05-02 (Actual)

PRIMARY OUTCOMES:
hospital acquired infections incidence | infections occured 48 hours after admission to ICU/PC-ICU
  cumulative incidence of bloodstream infections (BSI), central line-associates BSI (CLABSI), urinary tract infections (UTI), catheter-associated UTI (CAUTI) and ventilator-associated pneumonias (VAP)

SECONDARY OUTCOMES:
Ventilator-associated pnemonias (VAP) incidence | infections occured 48 hours after admission to ICU/PC-ICU
  VAP incidence
Bloodstream infections (BSI) incidence | infections occured 48 hours after admission to ICU/PC-ICU
  BSI incidence
central-line associated BSI (CLABSI) incidence | infections occured 48 hours after admission to ICU/PC-ICU
  CLABSI incidence
urinary tract infections (UTI) incidence | infections occured 48 hours after admission to ICU/PC-ICU
  UTI incidence
catheter associated UTI (CAUTI) incidence | infections occured 48 hours after admission to ICU/PC-ICU
  CAUTI incidence
4% CHG daily bathing safety | at discharge, approximately up to 10 days
  overall mortality in the treatment and control arm
4% CHG daily bathing-related adverse events | at discharge, approximately up to 10 days
  4% CHG daily bathing-related adverse events in the treatment arm compared to standard soap-related adverse events
time till infection | at discharge, approximately up to 10 days
  time between admission to ICU/PC-ICU and infection occurrence

CONTACTS AND LOCATIONS:
Overall Officials: franco baldelli, Professor, Study Chair — Infectious Diseases Clinical, University Hospital of Perugia, Perugia, Italy

REFERENCES:
- [Derived] Pallotto C, Fiorio M, De Angelis V, Ripoli A, Franciosini E, Quondam Girolamo L, Volpi F, Iorio P, Francisci D, Tascini C, Baldelli F. Daily bathing with 4% chlorhexidine gluconate in intensive care settings: a randomized controlled trial. Clin Microbiol Infect. 2019 Jun;25(6):705-710. doi: 10.1016/j.cmi.2018.09.012. Epub 2018 Sep 26. PMID 30267930

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-27): https://cdn.clinicaltrials.gov/large-docs/63/NCT03639363/Prot_SAP_000.pdf